CLINICAL TRIAL: NCT00450424
Title: Facilitating Informed Decisions for MSI Testing
Brief Title: Educational CD-ROM Compared With Standard Informed Consent for Patients With Colorectal Cancer or a Family History of Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CDR0000443988; 04827 (Other: Fox Chase Cancer Center); R01CA109332-05 (NIH)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Colorectal Cancer; Hereditary Non-polyposis Colon Cancer
Keywords: colon cancer; rectal cancer; hereditary non-polyposis colon cancer; recurrent colon cancer; stage I colon cancer; stage IIA colon cancer; stage IIB colon cancer; stage IIIA colon cancer; stage IIIB colon cancer; stage IIIC colon cancer; stage IVA colon cancer; stage IVB colon cancer; recurrent rectal cancer; stage I rectal cancer; stage IIA rectal cancer; stage IIB rectal cancer; stage IIC rectal cancer; stage IIIA rectal cancer; stage IIIB rectal cancer; stage IIIC rectal cancer; stage IVA rectal cancer; stage IVB rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis; Colonic Neoplasms; Rectal Neoplasms | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Counseling (No Intervention): Participants will be given one of two counseling interventions regarding MSI testing: standard counseling or a CD-ROM intervention.
  Interventions: Other: counseling intervention; Other: CD-ROM intervention

INTERVENTIONS:
Other: counseling intervention — Participants in the Counseling intervention will meet with the study health educator who will provide the participant with the standard MSI informed consent form and provide a brief, standardized explanation of the MSI test. At that time, the participant can ask any questions s/he wishes to ask. The patients will either sign (or not sign, if they do not consent to have the test, or wish to think further about the decision) after this discussion. Participants who have further questions will be referred to either the attending physician or the genetics counselor at each hospital site.
Other: CD-ROM intervention — Participants who are randomized to the CD-ROM condition will complete the baseline interview and then meet with the health educator who will provide the participant with the standard MSI consent form and provide a brief, standardized explanation of the MSI test. At that time, the participant can ask any questions s/he wishes to ask. Next, the participant will be provided with the CD-ROM to view on a laptop computer in the clinic. Participants will also be given a copy of the CD-ROM to take home and keep for future reference. The CD-ROM patients will sign (or not sign, if they do not consent or wish to think further about the decision) the consent form after this discussion.

SUMMARY:
RATIONALE: The use of a CD-ROM may help patients with colorectal cancer or a family history of colorectal cancer make informed decisions about undergoing microsatellite instability (MSI) testing.

PURPOSE: This randomized clinical trial is studying an educational CD-ROM to see how well it works compared with standard informed consent to assist decision-making about MSI testing in patients with colorectal cancer or a family history of colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the impact of standard informed consent vs a CD-ROM educational intervention on knowledge about microsatellite instability (MSI) testing in patients with colorectal cancer (CRC) or a family history of CRC.
* Determine the impact of these interventions on patient satisfaction with the preparation to make a decision.

Secondary

* Determine whether the CD-ROM educational intervention has a differential impact on satisfaction with the MSI test decision, difficulty making the MSI test decision, and decisional conflict, as well as on patients' attitudes about MSI testing and CRC (e.g., perceived benefits and barriers to having the MSI test, perceived risk for colorectal and related cancers, self-efficacy), on general and cancer-related distress, and on discussions with family members about the MSI test and familial CRC risk.
* Assess whether demographic factors, disease/family history characteristics, family support for testing, and cancer-related distress moderate the impact of the intervention on satisfaction with and completeness of the informed consent process.

OUTLINE: This is a multicenter, pilot, study (part I) followed by a randomized study (part II).

* Part I: The educational CD-ROM is developed over 9 months. Patients receive a pilot version of the CD-ROM and provide feedback regarding usability and content.
* Part II: Patients are randomized to 1 of 2 arms.

  * Arm I: Patients complete a baseline interview and receive a standard informed consent for microsatellite instability (MSI) testing and a brief, standardized explanation of the MSI test.
  * Arm II: Patients complete a baseline interview and receive a standard informed consent for MSI testing and the educational CD-ROM developed in phase I.

All patients in part II (even those that did not consent to the MSI test) complete a follow-up survey at 2 weeks.

Tissue samples from patients are analyzed by immunohistochemistry and MSI assay (polymerase chain reaction) for MLH1 and MSH2.

PROJECTED ACCRUAL: A total of 184 patients will be accrued for this study.

ELIGIBILITY:
Patient or family member meeting 1 of the following revised Bethesda colorectal cancer (CRC) criteria:

* Diagnosis of colon or rectal cancer at < 50 years of age
* Diagnosis of > 1 CRC at one time in the past
* Diagnosis of ≥ 1 CRC at different times
* Diagnosis of CRC and any other hereditary nonpolyposis colorectal cancer (HNPCC)-related cancers
* Diagnosis of CRC in ≥ 2 first-degree or second-degree relatives with HNPCC-related tumor and ≥ 1 cancer diagnosed at < 50 years of age
* Diagnosis of CRC in ≥ 2 first- or second-degree relatives with HNPCC-related tumors, regardless of age
* Diagnosis of CRC with pathologic features suggestive of microsatellite instability (MSI) and < 60 years of age

  * Patients with CRC meeting the Amsterdam criteria defined below are ineligible:
* Three relatives with CRC with 1 being a first-degree relative of the other 2
* Cases that span ≥ 2 generations
* At least 1 CRC case diagnosed before 50 years of age

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2007-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Manne, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (3):
- United States (3):
  - Helen F. Graham Cancer Center at Christiana Hospital, Newark, Delaware
  - Massachusetts General Hospital, Boston, Massachusetts
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Manne SL, Meropol NJ, Weinberg DS, Vig H, Ali-Khan Catts Z, Manning C, Ross E, Shannon K, Chung DC. Facilitating informed decisions regarding microsatellite instability testing among high-risk individuals diagnosed with colorectal cancer. J Clin Oncol. 2010 Mar 10;28(8):1366-72. doi: 10.1200/JCO.2009.25.0399. Epub 2010 Feb 8. PMID 20142594
- [Result] Hall MJ, Manne SL, Winkel G, Chung DS, Weinberg DS, Meropol NJ. Effects of a decision support intervention on decisional conflict associated with microsatellite instability testing. Cancer Epidemiol Biomarkers Prev. 2011 Feb;20(2):249-54. doi: 10.1158/1055-9965.EPI-10-0685. Epub 2011 Jan 6. PMID 21212064

RESULTS

PARTICIPANT FLOW:
Groups:
- CD-ROM Condition: Participants who are randomized to the CD-ROM condition will complete the baseline interview and then meet with the health educator who will provide the participant with the standard MSI consent form and provide a brief, standardized explanation of the MSI test. At that time, the participant can ask any questions s/he wishes to ask. Next, the participant will be provided with the CD-ROM to view on a laptop computer in the clinic. Participants will also be given a copy of the CD-ROM to take home and keep for future reference. The CD-ROM patients will sign (or not sign, if they do not consent or wish to think further about the decision) the consent form after this discussion.
- Standard Consent Condition: Participants in the Standard consent condition will complete the baseline interview and then meet with the study health educator who will provide the participant with the standard MSI informed consent form and provide a brief, standardized explanation of the MSI test. At that time, the participant can ask any questions s/he wishes to ask. The patients will either sign (or not sign, if they do not consent to have the test, or wish to think further about the decision) after this discussion. Participants who have further questions will be referred to either the attending physician or the genetics counselor.
Period: Overall Study
Arm/Group | CD-ROM Condition | Standard Consent Condition
Started | 122 | 117
Completed | 102 | 106
Not Completed | 20 | 11

BASELINE CHARACTERISTICS:
Groups:
- Standard Consent Condition: Participants in the Standard consent condition will complete the baseline interview and then meet with the study health educator who will provide the participant with the standard MSI informed consent form and provide a brief, standardized explanation of the MSI test. At that time, the participant can ask any questions s/he wishes to ask. The patients will either sign (or not sign, if they do not consent to have the test, or wish to think further about the decision) after this discussion. Participants who have further questions will be referred to either the attending physician or the genetics counselor at each hospital site.
- Total: Total of all reporting groups
Arm/Group | Standard Consent Condition | CD-ROM Condition | Total
Number analyzed (Participants) | 117 | 122 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.69 (7.38) | 47.33 (8.58) | 46.53 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 52 | 109
  Male | 60 | 70 | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 4 | 13
  White | 102 | 112 | 214
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 114 | 120 | 234
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Impact of Standard Informed Consent vs CD-ROM Educational Intervention on Knowledge About Microsatellite Instability (MSI) Testing
Description: 10-item true/false MSI knowledge survey developed by the oncologists on trial. (e.g., "Microsatellite Instability is found in every person that has had cancer."; "Microsatellite Instability may be caused by a permanent change in a gene that is inherited from a person's mother or father."). Participants can score anywhere from 0 (no questions answered correctly) to 10 (all questions answered correctly).
Time Frame: 2 weeks after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Consent Condition | CD-ROM Condition
Number analyzed (Participants) | 106 | 102
units on a scale | 4.07 (2.25) | 4.17 (2.94)

2. Secondary Outcome: Differential Impact of CD-ROM on Satisfaction With MSI Test Decision, Difficulty Making Decision & Decisional Conflict; Attitude; General & Cancer-related Distress; Discussions With Family About MSI Test & Familial Colorectal Cancer Risk
Description: Participants completed a baseline survey upon enrollment to the trial. 2 weeks after baseline, they completed a follow-up survey (assessed at both baseline and FU). Differential impact of CD-ROM on satisfaction with MSI test decision, difficulty making decision & decisional conflict; attitude; general & cancer-related distress; discussions with family about MSI test & familial colorectal cancer risk were measured.
Time Frame: at enrollment and 2 weeks after enrollment
Reporting Status: Not Posted

3. Secondary Outcome: Impact of Demographic Factors, Disease/Family History Characteristics, Family Support, and Cancer-related Distress on Satisfaction With and Completeness of the Informed Consent Process
Description: Participants completed a baseline survey upon enrollment to the trial. 2 weeks after baseline, they completed a follow-up survey (assessed at both baseline and FU). Impact of demographic factors, disease/family history characteristics, family support, and cancer-related distress on satisfaction with and completeness of the informed consent process was measured
Time Frame: at enrollment and 2 weeks after enrollment
Reporting Status: Not Posted

4. Secondary Outcome: Patient Satisfaction With the Preparation to Make a Decision
Description: Participants completed a baseline survey upon enrollment to the trial. 2 weeks after baseline, they completed a follow-up survey (assessed at both baseline and FU).
Time Frame: at enrollment and 2 weeks after enrollment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at baseline and follow up (2 weeks after baseline)
Description: Only adverse events related to emotional distress were collected. Participants will be asked at both survey time points about their emotional distress "how upset are you right now?" on a 7 point Likert scale. If the participant's rating is a 6 or a 7, an adverse event will be reported.
Arm/Group | Standard Consent Condition | CD-ROM Condition
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/122
Other Adverse Events (participants affected / at risk) | 0/117 | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No